CLINICAL TRIAL: NCT06322888
Title: Resistance and Aerobic Exercise for Prevention in Women With Dense Breasts (REP-D)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Jennifer A. Ligibel, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-676
Record Dates: First submitted 2024-03-01; First posted 2024-03-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Breast Cancer Female
Keywords: Breast Cancer; Breast Cancer Female; Breast Cancer Risk; Dense breast tissue; Dense breasts
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Exercise Intervention (Experimental): Participants will be randomized and will complete:
  * Baseline study visit with assessments, breast biopsy, and blood draw.
  * Exercise program for 12 weeks 3x weekly and exercise logs. Additional blood draw after first exercise session.
  * End of study visit with assessments, breast biopsy, and blood draw.
  Interventions: Behavioral: Exercise Training Program
- Arm B: Waitlist Control (No Intervention): Participants will be randomized and will complete:
  * Baseline study visit with assessments, breast biopsy, and blood draw.
  * End of study visit with assessments, breast biopsy, and blood draw.
  * Participants will be offered a complimentary 12-week exercise program after completing the study.

INTERVENTIONS:
Behavioral: Exercise Training Program — A 12-week aerobic and resistance-training exercise intervention with a certified exercise trainer in person or virtually. FitBit activity tracker, resistance bands, hand weights, and stationary bike will be provided to participants. Hand weights will be returned at end of study.
  Arms: Arm A: Exercise Intervention

SUMMARY:
The goal of this study is to learn more about how exercise might lower the risk of developing breast cancer in women with dense breast tissue by studying changes that occur in breast tissue and blood as a result of participating in an exercise program.

The names of the study groups in this study are:

* Exercise Training Group
* Waitlist Control Group

DETAILED DESCRIPTION:
The goal of this study is to learn more about how exercise might lower the risk of developing breast cancer by studying changes that occur in breast tissue and blood as a result of participating in an exercise program. Participants will be placed into one of two study groups: Exercise Training Group vs. Waitlist Control Group. Randomization means that a participant is put into a group by chance.

The research study procedures include screening for eligibility and baseline and end of study assessments which include: breast biopsies, assessment of physical activity habits, aerobic and strength testing, blood draws and questionnaires.

Participants randomized to the exercise group will be expected to participate in exercise sessions throughout the study. They will also be asked to complete logs of their activity.

Participants will be in this research study for up to 16 weeks.

It is expected that 46 women will take part in this study.

The Breast Cancer Research Foundation is supporting this research study by providing funding.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-59
* Heterogeneously dense/extremely dense (BIRADS 3 or 4) breast tissue on mammogram within the past 12 months
* Physically inactive; engaging in <60 minutes of moderate or vigorous intensity exercise per week, as assessed by Godin Leisure Time screener
* Not pregnant or breastfeeding
* English speaking and able to read English. Investigators are only enrolling English-speaking participants to this study at this time due to the fact that investigators currently only have English-speaking exercise trainers with the proper qualifications to conduct the exercise training
* Written informed consent prior to any study-related procedures

Exclusion Criteria:

* Self-reported inability to walk 2 blocks (at any pace)
* Prior history of breast cancer; prior DCIS is allowable as long as participant is not taking endocrine therapy and has at least 1 breast that has not been irradiated
* On oral or implantable hormonal contraceptives, postmenopausal hormone replacement therapy, a selective estrogen receptor modulator or an aromatase inhibitor; Mirena or other IUD is acceptable
* Consistent strength training in the past 3 months
* Use of weightloss drugs
* Cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate exercise. Examples would include unstable angina, recent myocardial infarction, oxygen-dependent pulmonary disease, and osteoarthritis requiring imminent joint replacement. Moderate arthritis that does not preclude physical activity is not a reason for ineligibility
* Psychiatric disorders or conditions that would preclude participation in the study intervention (e.g. untreated major depression or psychosis, substance abuse, severe personality disorder)

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 46 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Irisin in Exercise Group | At baseline, within 2 hours of 1st exercise session, and at week 12, up to 16 weeks
  Change in circulating irisin at baseline, after 1st exercise session, and end of study in exercise group, and it will be compared using Wilcoxon rank-sum testing. Irisin will be measured by Parallel Reaction Monitoring in the Spiegelman Lab, using the method described by Jedrychowski.
Change in Irisin in Control Group | At baseline and week 12, up to 16 weeks
  Change in circulating irisin at baseline and end of study in control group, and it will be compared using Wilcoxon rank-sum testing. Irisin will be measured by Parallel Reaction Monitoring in the Spiegelman Lab, using the method described by Jedrychowski.

SECONDARY OUTCOMES:
Change in Tissue Markers in Exercise Group | At baseline and week 12, up to 16 weeks
  Immunofluorescence analysis of immune and proliferative markers from biopsies of benign breast tissue will be assessed through C-detection by indexing (CODEX) imaging for the exercise group and will be compared between treatments using Wilcoxon rank-sum testing. Imaging to be performed by the Molecular Imaging Core (MIC) at Dana-Farber Cancer Institute.
Change in Tissue Markers in Control Group | At baseline and week 12, up to 16 weeks
  Immunofluorescence analysis of immune and proliferative markers from biopsies of benign breast tissue will be assessed through C-detection by indexing (CODEX) imaging for the exercise group and will be compared between treatments using Wilcoxon rank-sum testing. Imaging to be performed by the Molecular Imaging Core (MIC) at Dana-Farber Cancer Institute.
Change in Biomarkers in Exercise Group - Meso scale | At baseline and week 12, up to 16 weeks
  Assessed by assays for inflammatory mediators and will be performed using a Meso Scale Discovery multi-plex analysis system and will be conducted by the Translational Research Laboratory at Dana-Farber Cancer Institute.
Change in Biomarkers in Exercise Group - Mass cytometry | At baseline and week 12, up to 16 weeks
  Mass cytometry (CyTOF) will be used to evaluate a panel of immune mediators and will be performed in conjunction with the Polyak Laboratory. Wilcoxon rank-sum testing will be used to compare between treatments.
Change in Biomarkers in Control Group - Meso Scale | At baseline and week 12, up to 16 weeks
  Assessed by assays for inflammatory mediators and will be performed using a Meso Scale Discovery multi-plex analysis system and will be conducted by the Translational Research Laboratory at Dana-Farber Cancer Institute. Additionally, Mass cytometry (CyTOF) will be used to evaluate a panel of immune mediators and will be performed in conjunction with the Polyak Laboratory. Wilcoxon rank-sum testing will be used to compare between treatments.
Change in Biomarkers in Control Group - Mass cytometry | At baseline and week 12, up to 16 weeks
  Mass cytometry (CyTOF) will be used to evaluate a panel of immune mediators and will be performed in conjunction with the Polyak Laboratory. Wilcoxon rank-sum testing will be used to compare between treatments.
Change in Participant Weight in Exercise Group | At baseline and week 12, up to 16 weeks
  Defined as the percent change in weight for Exercise Group from pretreatment to week 12 will be calculated, summarized, and compared using Wilcoxon rank-sum testing.
Change in Participant Weight in Control Group | At baseline and week 12, up to 16 weeks
  Defined as the percent change in weight for Control Group from pretreatment to week 12 will be calculated, summarized, and compared using Wilcoxon rank-sum testing.
Change in Cardiorespiratory Fitness in Exercise Group | At baseline and week 12, up to 16 weeks
  Assessed by VO2 max (i.e., the number of milliliters of oxygen used per kilogram of body weight in one minute (ml/kg/min)), measured using the Sub-Maximal Cycle Ergometer Test, will be calculated and compared using Wilcoxon rank-sum testing.
Change in Cardiorespiratory Fitness in Control Group | At baseline and week 12, up to 16 weeks
  Assessed by VO2 max (i.e., the number of milliliters of oxygen used per kilogram of body weight in one minute (ml/kg/min)), measured using the Sub-Maximal Cycle Ergometer Test, will be calculated and compared using Wilcoxon rank-sum testing.
10-Repetition Max Test in Exercise Group | At baseline and week 12, up to 16 weeks
  The 10-Repetition Max Test is defined as the heaviest weight a participants could lift for 10 repetitions. Change and relative percent change will be calculated and compared between treatments using Wilcoxon rank-sum testing.
10-Repetition Max Test in Control Group | At baseline and week 12, up to 16 weeks
  The 10-Repetition Max Test is defined as the heaviest weight a participants could lift for 10 repetitions. Change and relative percent change will be calculated and compared between treatments using Wilcoxon rank-sum testing.
Change in Minutes of Total Exercise for Exercise Group | Up to 16 weeks
  Change in minutes of total exercise and met hours per week (7-day par) will be calculated and compared between treatments using Wilcoxon rank-sum testing. The proportion of participants that achieve 150 minutes of exercise per week by 12 weeks will be compared using Wilcoxon rank-sum testing and Fisher's exact tests.
Change in Minutes of Total Exercise for Control Group | Up to 16 weeks
  Change in minutes of total exercise and met hours per week (7-day par) will be calculated and compared between treatments using Wilcoxon rank-sum testing. The proportion of participants that achieve 150 minutes of exercise per week by 12 weeks will be compared using Wilcoxon rank-sum testing and Fisher's exact tests.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ligibel, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu